CLINICAL TRIAL: NCT04845919
Title: A Pilot Study to Evaluate the Safety and Feasibility of Sonodynamic Therapy Using the ExAblate MRI-Guided Focused Ultrasound in the Treatment of Cerebral Glioblastomas.
Brief Title: Sonodynamic Therapy with ExAblate System in Glioblastoma Patients
Acronym: Sonic ALA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Sonic ALA
Record Dates: First submitted 2021-04-02; First posted 2021-04-15 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Glioblastoma Multiforme
Keywords: Sonodynamic therapy,; focused ultrasound,; 5-aminolevulinic acid
MeSH Terms: conditions — Glioblastoma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 5-ALA mediated sonodynamic therapy (Experimental)
  Interventions: Drug: 5-Aminolevulinic Acid

INTERVENTIONS:
Drug: 5-Aminolevulinic Acid — SDT treatment with 5-ALA using the ExAblate Model 4000 Type-2 "Neuro-System".

SUMMARY:
The goal of this prospective, non-randomized, single-arm study is to evaluate the safety and feasibility of sonodynamic therapy with 5-aminolevulinic acid in patients with newly diagnosed cerebral glioblastomas using the ExAblate Model 4000 Type-2 "Neuro-System".

Patients will be consented, screened, and will undergo study SDT treatment with 5-ALA using the ExAblate Model 4000 Type-2 "Neuro-System". After SDT treatment, patients will perform a strict neuro-radiological follow-up (minimum of 2 MRI) and undergo tumor resection 15-21 days after SDT, according to the clinical and radiological status.

The main goal of the present study is to investigate the safety and feasibility of SDT in patients affected by GBMs attained with low-frequency FUS.

In particular:

Safety will be evaluated by patient examination and MRI images during the treatment, and by follow-up MRI and clinical and neurological visits.

To evaluate feasibility, the extent of the sonicated area will be calculated at the end of the procedure in order to evaluate the targeted area.

Secondary objective of the trial is to assess the efficacy of the SDT procedure in terms of tumor regression and/or cell apoptosis and necrosis.

DETAILED DESCRIPTION:
Despite progress made in many cancer treatments, High-Grade Gliomas (HGG) remain an extraordinary challenge. Their aggressive and infiltrative nature, the limited efficacy and inherent risk of surgical resection combined with radiotherapy, and the difficulty in delivering anticancer drugs to the brain, make the prognosis for patients with gliomas grim. Therefore, new and less-invasive alternatives to existing procedures are needed.

Sono-Dynamic Therapy (SDT) represents an emerging approach that offers the possibility of noninvasively eradicating solid tumors in a site-directed manner. It involves the delivery of a non-toxic chemical agent that selectively accumulates into target areas and the subsequent exposure of the targeted tissue to relatively low-intensity ultrasound. These procedures (sensitization and ultrasound exposure) are both per se harmless, but, when combined, result in activation of the chemical agent and subsequent cytotoxic events limited to the target tissue volume. SDT offers significant advantages because ultrasound energy can be tightly focused and delivered through the intact skull to deep areas of the brain, depending on the frequency. SDT is achieved by focusing low-intensity and lowfrequency ultrasound, which, as opposite to high-intensity ultrasonic beams, can be focused effectively within the whole intracranial space with the currently available device ExAblate 4000, Insightec, Haifa, Israel). This would enable to target also tumors in the peripheral area of the intracranial space. 5-ALA is a PpIX (Protoporphyrin IX) precursor that selectively accumulates in HGGs because of an enhanced uptake and metabolism from tumor cells. It is used for intra-operative guidance in surgery as tumoral tissues shows an exceeding fluorescence under certain light conditions due to PpIX accumulation, as compared to the normal surrounding parenchyma. It is therefore a good candidate for SDT. 5-ALA can exert sono-dynamic effects against HGGs, as it has been shown in several preclinical studies. Pre-clinical data on a safety experiment conducted at the University of Virginia showed that SDT with 5-ALA was not exerting a toxic effect to the normal brain [Raspagliesi L. et al. 2021].

The idea of the present study is to investigate the antitumor effects of SDT in patients affected by HGGs attained with low-frequency Focused Ultrasound. Focused Ultrasound under MRI-guidance can be safely delivered through an intact human skull to perform SDT in combination with 5-ALA with a low risk of transient adverse effects, and will be evaluated during follow-up visits, postprocedural serial MRI, and histology.

The main goal of this prospective, non-randomized, single-arm study is to evaluate the safety and feasibility of SDT in patients with newly diagnosed cerebral glioblastomas using the ExAblate Model 4000 Type-2 "Neuro-System". The ExAblate Model 4000 Type-2 "Neuro-System" is intended for use as a tool to induce targeted tumor's inhibition of growth and cell destruction in patients with cerebral lobar glioblastomas.

Patients harboring newly diagnosed lobar glioblastoma according to RANO criteria will provide informed consent, will be screened, and will undergo study SDT treatment using the ExAblate Model 4000 Type-2 "Neuro-System". After SDT treatment, patients will perform a strict neuro-radiological follow-up (minimum of 2 MRI) and undergo tumor resection about 15-21 days after SDT, according to the clinical and radiological status.

The main purpose of this study is to evaluate the safety and feasibility of SDT. In particular, safety will be evaluated by patient examination and MRI during the treatment, and by follow-up by daily clinical visits and MRI every 5 (± 2) days according to clinical and radiologic findings. Safety data will be assessed during each visit through a combination of MRI evaluations, clinical assessments, and neurological examinations, according to the clinical findings assessed until the decision to proceed with surgical resection. Feasibility will be evaluated performing 4 MRI (Day 1, 5, 10, 15) after SDT treatment evaluating tumor size, morphology and perilesional edema until tumor resection.

A secondary objective of the present study is to assess the efficacy of the treatment; in particular, to investigate the antitumor effects of SDT in patients affected by HGGs attained with low-frequency

Focused Ultrasound, the following data will be collected:

* Tumor volume changes after SDT according to sonicated tumors volumes (by imaging).
* Histology after tumor resection, comprising assessment of apoptosis and necrosis.

Despite all current treatment modalities, glioblastoma patient's prognosis remains dismal. By proving that procedure is safe and feasible this study will establish the SDT treatment modality as a possible alternative or a synergistic tool to current treatment modalities. It will also pave the way to the application of SDT in other forms of brain tumors, both intra- and extra-axial, and to the development of tumor specific sono-sensitizers.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, age between 18 and 75 years, inclusive.
2. Suspected primary lobar Glioblastoma clearly measurable on the basis of Response Assessment in Neuro-Oncology (RANO) criteria
3. Newly diagnosed brain glioblastomas located in a surgically accessible brain region for resection
4. The targeted tumor resection volume measures between 1 cm and 6 cm in diameter.
5. Karnofsky rating 70-100.
6. ASA score 1-3.
7. Able to attend all study visits.
8. No previous brain surgery.
9. No previous radiation treatment.
10. No previous systemic treatment for the tumor.
11. Able and willing to give Informed Consent.
12. No contraindication to MRI.
13. No contraindication to brain surgery.
14. Contraceptive use by both male and female subjects consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

    * Male participants: Male participants must agree that, if their partner is at risk of becoming pregnant, they will use an effective method of contraception. The participants must agree to use the contraception during the whole period of the study and for 12 weeks after the study intervention injection.
    * Female participants: A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies: (i) is a woman of nonchildbearing potential (WONCBP) as defined in Appendix C Contraception and Barrier Guidance OR (ii) is a WOCBP and using an acceptable contraceptive method as described in Appendix C: Contraceptive and Barrier Guidance during the study intervention period (at a minimum until after the last dose of study intervention).

Exclusion Criteria:

1. Brain glioblastoma presenting with the following characteristics:

   * Brain edema and/or mass effect that causes midline shift of more than 15 mm
   * Evidence of recent intracranial hemorrhage within the targeted tumor volume
   * Calcifications in the focused ultrasound sonication path (system tools may not tailor the treatment around these calcifications)
2. The sonication pathway to the tumor involves either:

   * more than 30% of the skull area traversed by scars, scalp disorders (e.g., eczema), or atrophy of the scalp
   * Clips, shunts, or other metallic implanted objects in the skull or the brain
3. Cardiac disease or unstable hemodynamic status including:

   * Documented myocardial infarction within six months of enrolment
   * Unstable angina on medication
   * Congestive heart failure
   * Left ventricular ejection fraction < 50%
   * Right-to-left, bidirectional, or transient right-to-left cardiac shunts
   * History of a hemodynamically unstable cardiac arrhythmia
   * Cardiac pacemaker
4. Severe hypertension
5. Anti-coagulant therapy or medications known to increase risk of hemorrhage within washout period prior to treatment
6. History of a bleeding disorder, coagulopathy or with a history of spontaneous tumor hemorrhage
7. Abnormal level of platelets (<100000) or INR >1.3
8. Cerebral or systemic vasculopathy
9. Known allergy sensitivity or contraindications to gadolinium
10. Contraindications to MRI such as non-MRI-compatible implanted devices
11. Subjects not fitting comfortably into the MRI scanner
12. Difficulty lying supine and still for up to 4 hours in the MRI unit or claustrophobia
13. Positive pregnancy test (for pre-menopausal women) (see Appendix C)
14. Severely impaired renal function with estimated glomerular filtration rate <30mL/min/1.73m2 and/or on dialysis
15. Respiratory: chronic pulmonary disorders (e.g., severe emphysema, COPD, pulmonary vasculitis, or other causes of reduced pulmonary vascular cross-sectional area).
16. Other contraindications to 5-ALA, including chronic or acute porfiria, and hypersensibility to 5-ALA or porfirins
17. Any illness or medical condition that in the investigator's opinion precludes participation in this study
18. Patients unable to sign an Informed Consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Presence of hemorrhage, edema or other damages | 10 days after the procedure
  MR images will be acquired before the procedure and will also be used to guide the FUS treatment; new MRI scans will be acquired at immediately after and at 24 hours, 5 days and 10 days after the procedure and will be analyzed to identify any focal alteration within the treatment's radius compatible with hemorrhages, necrosis, oedema, inflammation or other damages

SECONDARY OUTCOMES:
Rate of neurological deficits | 10 days after the procedure
  Patients will be clinically evaluated to identify any change in their clinical picture or new onset of neurological symptoms/deficits,
Radiological response to treatment | 10 days after the procedure
  Tumor volume at baseline will be assessed for each patient as gadolinium-enhancing parenchymal regions before any follow-up scan. Post-treatment tumor volumes will be assessed at all follow-up MRI scans, and radiological response to sonodynamic therapy -i.e. the change in pathological volume after the treatment- will be determined by confronting baseline and follow-up scans by the RANO Criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation IRCCS Carlo Besta Neurological Institute, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonosi L, Marino S, Benigno UE, Musso S, Buscemi F, Giardina K, Gerardi R, Brunasso L, Costanzo R, Iacopino DG, Maugeri R. Sonodynamic therapy and magnetic resonance-guided focused ultrasound: new therapeutic strategy in glioblastoma. J Neurooncol. 2023 May;163(1):219-238. doi: 10.1007/s11060-023-04333-3. Epub 2023 May 14. PMID 37179515
- [Background] Pellegatta S, Corradino N, Zingarelli M, Porto E, Gionso M, Berlendis A, Durando G, Maffezzini M, Musio S, Aquino D, DiMeco F, Prada F. The Immunomodulatory Effects of Fluorescein-Mediated Sonodynamic Treatment Lead to Systemic and Intratumoral Depletion of Myeloid-Derived Suppressor Cells in a Preclinical Malignant Glioma Model. Cancers (Basel). 2024 Feb 15;16(4):792. doi: 10.3390/cancers16040792. PMID 38398183
- [Background] Keating GF, Chesney KM, Patel N, Kilburn L, Fonseca A, Packer RJ, Challa C, O'Brien PF, Donoho DA, Myseros JS, Oluigbo C, Keating RF, Syed HR. MR-guided focused ultrasound in pediatric neurosurgery: current insights, technical challenges, and lessons learned from 45 treatments at Children's National Hospital. Neurosurg Focus. 2024 Sep 1;57(3):E6. doi: 10.3171/2024.6.FOCUS24332. PMID 39217632
- [Background] Huangfu L, Zha B, Li P, Wang L, Liu X, Cui H, Li Y, Wu J, Shi S, Yang Y, Sun X, Gao S, Li H, Yang D, Zheng Y. A phase I clinical trial of sonodynamic therapy combined with radiotherapy for brainstem gliomas. Int J Cancer. 2025 Mar 1;156(5):1005-1014. doi: 10.1002/ijc.35218. Epub 2024 Oct 8. PMID 39377640